CLINICAL TRIAL: NCT05419869
Title: An Open-Label Study of ALTO-100 in Adults With Major Depressive Disorder (MDD)
Brief Title: Pilot Decentralized Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alto Neuroscience (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALTO-100-003
Record Dates: First submitted 2022-05-16; First posted 2022-06-15 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ALTO-100 (Experimental): ALTO-100 tablet PO ; twice daily dosing 8 weeks
  Interventions: Drug: ALTO-100 PO Tablet

INTERVENTIONS:
Drug: ALTO-100 PO Tablet — Two tablets daily

SUMMARY:
The purpose of this study is to collect biologically-based data for defining predictors and correlates of the effects of ALTO-100.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of moderate to severe major depressive disorder
* Either currently taking a SSRI, SNRI, mirtazapine, or bupropion for at least 6 weeks with no dose modifications in the past 2 weeks, or are not taking an antidepressant medication
* Willing to comply with all study assessments and procedures
* Must not be pregnant or breastfeeding at time of enrollment or throughout study
* Must have access with privacy to a computer with a keyboard and internet

Exclusion Criteria:

* Evidence of acute or unstable cardiovascular, respiratory, hepatic, or other major disease
* Active suicidal ideation
* Severe impediment to vision, hearing, and/or hand movement
* Diagnosed bipolar disorder or psychotic disorder
* Has a history of hypersensitivity or allergic reaction to ALTO-100 or any of its components/excipients
* Concurrent or recent participation in another clinical trial for mental illness involving an investigational product or device

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-01-13 (Actual); Study Completion 2023-01-26 (Actual)

PRIMARY OUTCOMES:
To understand the relationship between baseline biology and score change in the Montgomery-Asberg Depression Rating Scale (MADRS) with ALTO-100 from start of dosing to end of treatment | Measured at Day 1, Day 14, Day 28, Day 42, Day 56
  The Montgomery-Åsberg Depression Rating Scale (MADRS) measures the severity of depression where smaller scores indicate less depression and higher scores suggest more severe depression. Possible scores for this 10 item version range from 0 to 60. The score change from the start of dosing (Day 1) to the end of treatment (Day 56) is the primary outcome.
To understand the relationship between baseline biology and score change in the Clinical Global Impression scale - Severity (CGI-S) with ALTO-100 from Screening to end of treatment | Measured at Screening, Day 1, Day 14, Day 28, Day 42, Day 56
  The Clinical Global Impression scale - Severity (CGI-S) measures the severity of psychopathology in general where smaller scores indicate less illness and higher scores suggest more severe illness. Possible scores for this scale range from 1 to 7. The score change from Screening (Day [-21]) to the end of treatment (Day 56) is the primary outcome.
Number of Participants with Adverse Events (AEs) as a Measure of Safety and Tolerability of ALTO-100 | From the signing of the ICF until the follow-up visit (up to 13 weeks)
  An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.
Number of Participants With Clinically Significant Laboratory Abnormalities as a Measure of Safety and Tolerability of ALTO-100 | From the signing of the ICF until the end-of-treatment visit (up to 13 weeks)
  Blood samples for serum chemistry and hematology will be collected for clinical laboratory testing.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Site 160, Coral Gables, Florida
  - Site 156, Jackson, Mississippi